CLINICAL TRIAL: NCT01771107
Title: A Pilot Trial of AVD and Brentuximab Vedotin (SGN-35) in the Treatment of Stage II-IV HIV-Associated Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Combination Chemotherapy in Treating Patients With Stage II-IV HIV-Associated Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00046; NCI-2013-00046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-003678-18; 085; AMC-085 (Other: AIDS Malignancy Consortium); AMC-085 (Other: CTEP); UM1CA121947 (NIH); NCT02298257 (obsolete NCT alias)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: AIDS-Related Hodgkin Lymphoma; Ann Arbor Stage II Hodgkin Lymphoma; Ann Arbor Stage IIA Hodgkin Lymphoma; Ann Arbor Stage IIB Hodgkin Lymphoma; Ann Arbor Stage III Hodgkin Lymphoma; Ann Arbor Stage IIIA Hodgkin Lymphoma; Ann Arbor Stage IIIB Hodgkin Lymphoma; Ann Arbor Stage IV Hodgkin Lymphoma; Ann Arbor Stage IVA Hodgkin Lymphoma; Ann Arbor Stage IVB Hodgkin Lymphoma; Classic Hodgkin Lymphoma; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Brentuximab Vedotin; Dacarbazine; Doxorubicin; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (brentuximab and combination chemotherapy) (Experimental): Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Pharmacological Study; Drug: Vinblastine

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Pharmacological Study — Correlative studies
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB

SUMMARY:
This pilot phase I/II trial studies the side effects and the best dose of brentuximab vedotin when given together with combination chemotherapy and to see how well they work in treating patients with stage II-IV human immunodeficiency virus (HIV)-associated Hodgkin lymphoma. Brentuximab vedotin is a monoclonal antibody, called brentuximab, linked to a chemotherapy drug called vedotin. Brentuximab attaches to CD30-positive cancer cells in a targeted way and delivers vedotin to kill them. Drugs used in chemotherapy, such as doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving brentuximab vedotin together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To identify the maximum tolerated dose (MTD) of brentuximab vedotin when combined with the doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine (AVD) chemotherapy regimen in the treatment of HIV-associated stage II-IV Hodgkin lymphoma. (Phase I) II. Establish an estimate of the two-year progression-free survival (PFS) for participants with HIV-associated stage II-IV Hodgkin lymphoma when treated using brentuximab vedotin plus the AVD chemotherapy regimen. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of AVD and brentuximab vedotin with highly active antiretroviral therapy (HAART).

II. To estimate the partial response (PR) rate, complete response (CR) rate, overall survival (OS), and event free survival (EFS) at 2 and 5 years.

III. To evaluate the effect of AVD and brentuximab vedotin on cluster of differentiation (CD)4 and CD8 counts after cycle 1, 4, at the end of therapy, and every 3 months after treatment completion for one year.

IV. To investigate the prognostic value of fludeoxyglucose (FDG)-positron emission tomography (PET)/computed tomography (CT) scans at baseline, after cycle 2, and at treatment completion, with respect to 2-year progression free survival.

V. To evaluate HAART status at baseline and to correlate this with tumor response to therapy and OS and PFS.

VI. To characterize the histologic subtypes in HIV-Hodgkin lymphoma (HL) in the highly active antiretroviral therapy (HAART) era.

VII. To assess the neurotoxicity of HAART in combination with AVD and brentuximab vedotin.

VIII. To evaluate effect of AVD and brentuximab vedotin on viral load after cycles 1, 4, at the completion of therapy, and every 3 months after treatment completion for one year.

IX. To perform pharmacokinetic and immunogenicity studies to determine drug levels during therapy.

X. To perform micro ribonucleic acid (miRNA) profile analysis on the HIV-HL tumor specimens and to correlate miRNA expression with OS, PFS, tumor response to therapy, histologic subtype of HIV-HL, and HIV disease characteristics.

XI. To perform tissue microarray analysis on HIV-HL tumor specimens and to correlate the markers studied with OS, PFS, and tumor response to therapy.

XII. To identify Epstein-Barr virus (EBV)-associated tumor derived deoxyribonucleic acid (DNA) in the plasma of study participants and to correlate these levels during therapy with disease response and OS. (Phase II) XIII. To identify cytokines in the plasma of participants during therapy that can be used as tumor and prognostic markers. (Phase II) XIV. To assess latent and expressed HIV reservoirs before, during, and post chemotherapy. To understand how cytotoxic chemotherapeutic agents affect HIV expression.

OUTLINE: This is a phase I, dose-escalation study of brentuximab vedotin followed by a phase II study.

Patients receive doxorubicin hydrochloride intravenously (IV), vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive; documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care provider;
  * Documentation of receipt of antiretroviral therapy (ART) by a licensed health care provider;
  * HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating > 1000 RNA copies/mL;
  * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 western blot confirmation or HIV rapid multispot antibody differentiation assay
  * NOTE: A "licensed" assay refers to a United States (US) Food and Drug Administration (FDA)-approved assay, which is required for all investigational new drug (IND) studies
* Histologic diagnosis of CD30-positive classical HL as defined by the 2008 World Health Organization (WHO) Classification of Hematological diseases; nodular lymphocyte predominant Hodgkin lymphoma is not eligible
* Stage II, III or IV disease as defined by the Ann Arbor Staging System
* Participants must have previously untreated HIV-classical HL (cHL), with the exception of up to 14 consecutive days of steroids, emergency radiation, or 1 prior cycle of cyclophosphamide to reduce tumor burden and improve hyperbilirubinemia in the setting of lymphoma related liver involvement
* Normal baseline cardiac ejection fraction >= 50%
* Serum creatinine of =< 1.5 mg/dL; if creatinine > 1.5 mg/dL, creatinine clearance must be >= 60 mL/minute
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 75,000/uL unless related to bone marrow involvement by HIV-cHL
* Total bilirubin must be < 1.5 x the upper limit of normal, unless the elevation of bilirubin is thought to be secondary to Gilbert's syndrome or combined antiretroviral therapy (cART); if, however, the elevated bilirubin is felt to be secondary to antiretroviral therapy, the total bilirubin must be =< 3.5 mg/dL, provided that the direct bilirubin is normal and the aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x the upper limit of normal; also, if the elevated bilirubin is thought to be secondary to cHL the same criteria for hyperbilirubinemia should be applied; however 1 prior cycle of cyclophosphamide is permitted in attempt to make the participant eligible; patients should not be excluded from study participation unless dosing cannot be safely established
* Female participants must have a negative pregnancy test within 1 week of enrollment and all participants must agree to use two reliable methods of contraception simultaneously if conception is possible during the study and for 6 months after stopping treatment; should a woman subject become pregnant or suspect she is pregnant while the subject is participating in this study, she should inform her treating physician immediately; the participant will then be removed from protocol therapy; participants who father a child while participating in the study will be permitted to continue with the protocol; the participant, however, is required to notify the investigator if he fathers a child
* Ability to understand and the willingness to sign a written informed consent document
* Karnofsky performance status > 30% (given the aggressiveness of this disease and the often severely debilitated nature of the patients at initial presentation)
* Measurable or non-measurable (evaluable) tumor parameter(s); non-measurable tumor parameters will be defined as not having bi-dimensional measurements (i.e., gastric or marrow involvement) but can be followed for response by other diagnostic tests such as gallium, PET imaging and/or bone marrow biopsy
* Patients already receiving erythropoietin or granulocyte colony stimulating factor (GCSF) for treatment of HIV-related cytopenia are eligible
* CD4 count >= 50 cells/ul
* Participants are required to be on antiretroviral regimens that are in accordance with the current International Acquired Immune Deficiency Syndrome (AIDS) Society guidelines concurrently with chemotherapy; the specific agents are at the discretion of the investigator and the use of investigational agents currently available on an expanded access basis is allowed; use of experimental antiretroviral agents or those containing zidovudine (including Combivir and Trizivir) or ritonavir (includes Norvir or Kaletra), cobicistat, didanosine (Videx or Videx EC), or similar potent cytochrome P450 (CYP)3 inhibitors are prohibited; in order to be eligible, participants taking zidovudine or ritonavir, or cobicistat, didanosine, or other CYP3 inhibitors must change to a different regimen 7 days prior to therapy initiation; changes to HAART therapy during the study may be made if medically necessary (toxicity, failure of regimen, etc.); participants must be on HAART at least 7 days prior to therapy
* Negative for hepatitis B, or if infected with hepatitis B, receiving anti-hepatitis B therapy; all participants will be required to be screened for hepatitis B; per Infectious Disease Society of America (IDSA) and Assistance for AIDS Specific Drugs (AASD) guidelines, those participants that show no immunity, defined by the lack of hepatitis B surface antigen antibody, and show evidence of chronic infection (i.e. hepatitis B surface antigen [HBsAg]+, hepatitis B core [HBcore]+, hepatitis B surface antibody [HBsAB]-) will be required to be on anti-hepatitis B therapy during the study in order to be eligible; patients will be permitted to enroll in the study provided normal liver function tests and no evidence of cirrhosis; the exact hepatitis B therapy will be at the discretion of the infection disease specialist or investigator; however all patients who present with acute hepatitis B or show normal transaminases and are hepatitis B virus HBsAg surface protein antigen (HBsAg) positive (+) and immunoglobulin M (IgM)+ for hepatitis core antigen will not be eligible for trial enrollment
* Patients diagnosed with hepatitis C who are hepatitis C antibody positive, whether hepatitis C RNA level is measurable or not, must have no evidence of cirrhosis and have liver function tests
* Brentuximab vedotin is partially metabolized via the CYP3A4 pathway and is cleared from the cells via the P-glycoprotein pump; therefore, participants must discontinue use of the following agents within 7 days prior to therapy

  * Strong CYP3A4 inhibitors that treat HIV
  * Other strong CYP3A inhibitors
  * Moderate CYP3A4 inhibitors should be used with caution but are not excluded; if 2 moderate CYP3A4 inhibitors are used concurrently, one must be discontinued at least 7 days (1 week) prior to the initiation of chemotherapy
  * P-glycoprotein inhibitors
  * If patients are taking any of these excluded medications, they must be discontinued at least 7 days (1 week) prior to the initiation of chemotherapy All concomitant medications must be reviewed by the study chair or co-chair prior to enrollment by email; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of

Exclusion Criteria:

* Patients with prior anthracycline therapy will be excluded
* Female participants who are pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta (b)-human chorionic gonadotropin (b-hCG) or urine pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Medical illness unrelated to HL, which in the opinion of the study physician will preclude administration of chemotherapy safely; this includes patients with uncontrolled infection (including opportunistic), chronic renal failure, myocardial infarction (MI) within the past 6 months, unstable angina, or cardiac arrhythmias other than chronic atrial fibrillation, or second malignancy requiring active treatment
* Prior malignancy within 2 years before enrollment other than curatively treated cutaneous basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, anal intraepithelial neoplasia, or cutaneous Kaposi's sarcoma (KS); participants with prior malignancies must have completed all therapy at least 2 years before enrollment with no evidence of disease since therapy completion
* Grade 2 or greater peripheral neuropathy
* Evidence of progressive multifocal leukoencephalopathy (PML) identified on the pretreatment magnetic resonance imaging (MRI)
* Central nervous system disease
* Patients with history of John Cunningham (JC) virus identified in the cerebrospinal fluid (CSF) or previous history of PML will be excluded from the study
* Cirrhosis secondary to any cause will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Rubinstein, Principal Investigator — AIDS Malignancy Consortium
Locations (28):
- United States (20):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University - Jewish, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- France (8):
  - Centre Hospitalier Universitaire (CHU) de Toulouse, Cedex
  - Hopital Antoine Beclere, Clamart
  - Henri Mondor University-Hospital Center, Créteil
  - Hopital l'Archet-CHU de Nice, Nice
  - Hopital Saint Louis, Paris
  - Hospital Saint-Antoine, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Chu Purpan, Toulouse

REFERENCES:
- [Derived] Rubinstein PG, Moore PC, Bimali M, Lee JY, Rudek MA, Chadburn A, Ratner L, Henry DH, Cesarman E, DeMarco CE, Costagliola D, Taoufik Y, Ramos JC, Sharon E, Reid EG, Ambinder RF, Mitsuyasu R, Mounier N, Besson C, Noy A; AIDS Malignancy Consortium; Lymphoma Study Association. Brentuximab vedotin with AVD for stage II-IV HIV-related Hodgkin lymphoma (AMC 085): phase 2 results from an open-label, single arm, multicentre phase 1/2 trial. Lancet Haematol. 2023 Aug;10(8):e624-e632. doi: 10.1016/S2352-3026(23)00157-6. PMID 37532416
- [Derived] Rubinstein PG, Moore PC, Rudek MA, Henry DH, Ramos JC, Ratner L, Reid E, Sharon E, Noy A; AIDS Malignancy Consortium (AMC). Brentuximab vedotin with AVD shows safety, in the absence of strong CYP3A4 inhibitors, in newly diagnosed HIV-associated Hodgkin lymphoma. AIDS. 2018 Mar 13;32(5):605-611. doi: 10.1097/QAD.0000000000001729. PMID 29280762

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Brentuximab 1.2 mg/kg: Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV
  Dacarbazine: Given IV
  Doxorubicin Hydrochloride: Given IV
  Pharmacological Study: Correlative studies
  Vinblastine: Given IV
- Phase II - Brentuximab 1.2 m/kg: Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV
Period: Overall Study
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Started | 6 | 35
Completed | 5 | 27
Not Completed | 1 | 8
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — participant moved | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participant enrolled on the study
Groups:
- Phase II - Brentuximab 1.2 mg/kg: Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV
  Dacarbazine: Given IV
  Doxorubicin Hydrochloride: Given IV
  Pharmacological Study: Correlative studies
  Vinblastine: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg | Total
Number analyzed (Participants) | 6 | 35 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (12.2) | 44.3 (12.0) | 43.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 33 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 9
  Not Hispanic or Latino | 5 | 16 | 21
  Unknown or Not Reported | 1 | 10 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 10 | 11
  White | 4 | 14 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 11 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 26 | 32
  France | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose of Brentuximab Vedotin (Phase I)
Description: Defined as the dose level at which =< 1 of 6 subjects experience dose limiting toxicity.
Time Frame: 28 days
Population: Participants entered into the phase I portion of the study
Measure: Number; unit: mg/kg
Arm/Group | Treatment (Brentuximab and Combination Chemotherapy)
Number analyzed (Participants) | 6
mg/kg | 1.2

2. Primary Outcome: 2-year Progression-free Survival (PFS) (Phase II)
Description: 2-year PFS is determined based on the Kaplan-Meier estimates and corresponding 95% confidence intervals based on standard errors using Greenwood's formula.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
proportion of participants | 1.0 [1.0 to 1.0] | 0.878 [0.706 to 0.953]

3. Secondary Outcome: Frequency of Adverse Events
Description: Number of Participants who had one or more adverse events
Time Frame: Up to 5 years
Population: Participants who were treated with brentuximab and combination chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
Participants | 6 | 35

4. Secondary Outcome: Partial Response Rate
Description: Number of participants who achieved a partial response per RECIST v1.0 criteria
Time Frame: 2 years
Population: Patients who completed therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
Participants | 1 | 4

5. Secondary Outcome: Partial Response Rate
Description: Number of participants who achieved a partial response per RECIST v1.0 criteria
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
Participants | 0 | 0

6. Secondary Outcome: Complete Response Rate
Description: Number of participants who experienced a complete response per RECIST v1.0 criteria
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
Participants | 6 | 32

7. Secondary Outcome: Complete Response Rate
Description: Number of participants who achieved a complete response per RECIST v1.0 criteria
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
Participants | 6 | 33

8. Secondary Outcome: 2-year Overall Survival
Description: Proportion of study participants who are alive at 2 years estimated using the Kaplan-Meier survival function
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
proportion of participants | 1.0 [1.0 to 1.0] | 0.91 [0.74 to 0.97]

9. Secondary Outcome: Overall Survival
Description: Proportion of participants who are alive at 5 years using a Kaplan-Meier estimate
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
proportion of participants | 1.0 [1.0 to 1.0] | 0.876 [0.7 to 0.952]

10. Secondary Outcome: Event-free Survival
Description: Proportion of participants who are alive and progression-free at 2 years
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Phase II Brentuximab 1.2 mg/kg: Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV on days 1 and 15. Patients also receive brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV
  Dacarbazine: Given IV
  Doxorubicin Hydrochloride: Given IV
  Pharmacological Study: Correlative studies
  Vinblastine: Given IV
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
proportion of participants | 1.0 [1.0 to 1.0] | 0.878 [0.706 to 0.953]

11. Secondary Outcome: Event-free Survival
Description: Binomial probabilities and their 95% confidence intervals will be used to estimate the response rates (i.e., partial response rate, complete response rate, overall response rate) and event free survival at 2 and 5 years of AVD and brentuximab vedotin for a treatment of patients with stage III/IV HIV-associated Hodgkin lymphoma.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
proportion of participants | 1.0 [1.0 to 1.0] | 0.743 [0.55 to 0.863]

12. Secondary Outcome: CD4 Counts
Description: CD4 counts (absolute) at visit 4 (cycle 5)
Time Frame: 5 months
Population: Participants with absolute cd4 counts at cycle 5
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 26
cells/µL | 378 [289 to 530] | 401 [292 to 481]

13. Secondary Outcome: CD8 Counts
Description: Absolute CD8 counts at cycle 5
Time Frame: 5 months
Population: Participants with absolute CD8 counts at cycle 5
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 26
cells/µL | 719.5 [596 to 883] | 666.5 [470 to 954]

14. Secondary Outcome: Viral Load
Description: HIV viral load (detectable)
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 5 | 27
Participants | 1 | 7

15. Secondary Outcome: Prognostic Value of Fludeoxyglucose F-18 (FDG)-Positron Emission Tomography (PET) in Patient With HIV and Hodgkin Lymphoma (HL) With Respect to 2 Year Progression Free Survival
Description: Log-rank analysis will be used to investigate the prognostic value of FDG-PET scans at baseline, after 2 courses and post-therapy in patients with HIV and HL with respect to progression free survival.
Time Frame: Baseline up to 2 years
Population: PET-CT positive status was used within each arm.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
proportion of participants
  PET-CT positive: number analyzed (Participants) | 6 | 33
  PET-CT positive | 0.876 [0.701 to 0.951] | 0.876 [0.701 to 0.951]
  PET-CT negative: number analyzed (Participants) | 0 | 2
  PET-CT negative |  | 0 [0 to 0]

16. Secondary Outcome: Prognostic Value of FDG-PET in Patient With HIV and HL With Respect to 2 Year Progression Free Survival
Description: as for outcome 15
Time Frame: Baseline up to 2 years
Population: PET-CT positive status was used within each arm.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 32
proportion of participants
  PET-CT positive: number analyzed (Participants) | 1 | 1
  PET-CT positive | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  PET-CT negative: number analyzed (Participants) | 5 | 31
  PET-CT negative | 1.0 [1.0 to 1.0] | 0.897 [0.714 to 0.966]

17. Secondary Outcome: Prognostic Value of FDG-PET in Patient With HIV and HL With Respect to 2 Year Progression Free Survival
Description: as for outcome 15
Time Frame: Baseline up to 2 years
Population: PET-CT positive status was used within each arm.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 5 | 28
proportion of participants
  PET-CT positive: number analyzed (Participants) | 0 | 2
  PET-CT positive |  | 1.0 [1.0 to 1.0]
  PET-CT negative: number analyzed (Participants) | 5 | 26
  PET-CT negative | 1.0 [1.0 to 1.0] | 0.92 [0.716 to 0.979]

18. Secondary Outcome: HAART Status
Description: Log-rank analysis will be used to evaluate HAART status at baseline for difference in outcome in terms of progression free survival at 2 years.
Time Frame: Baseline up to 2 years
Population: All participants had HAART at baseline. Logrank test cannot be performed.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
proportion of participants
  HAART yes | 1.0 [1.0 to 1.0] | 0.878 [0.706 to 0.953]
  HAART no: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: HAART Status
Description: Log-rank analysis will be used to evaluate HAART status at baseline for difference in outcome in terms of overall survival at 2 years.
Time Frame: Baseline up to 2 years
Population: All participant had HAART at baseline. Logrank test cannot be performed.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 m/kg
Number analyzed (Participants) | 6 | 35
proportion of participants
  HAART yes | 1.0 [1.0 to 1.0] | 0.911 [0.747 to 0.97]
  HAART no: number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Characterization of Histologic Subtypes in HIV-HL in the HAART Era
Description: Participants with mixed cellularity histologic subtype in HIV-HL in the HAART era
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 6 | 35
Participants | 2 | 13

21. Secondary Outcome: Incidence of Neurotoxicity
Description: Number of participants who experience neurotoxicity at cycle 5 (visit 4)
Time Frame: 5 months
Population: Participants who had neurotoxicity evaluated at cycle 5
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
Number analyzed (Participants) | 4 | 26
Participants | 4 | 23

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Phase I - Brentuximab 1.2 mg/kg | Phase II - Brentuximab 1.2 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 3/35
Serious Adverse Events (participants affected / at risk) | 3/6 | 16/35
Other Adverse Events (participants affected / at risk) | 6/6 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Brentuximab 1.2 mg/kg (N=6) | Phase II - Brentuximab 1.2 mg/kg (N=35)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Coronary artery disease (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Death, NOS (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Brentuximab 1.2 mg/kg (N=6) | Phase II - Brentuximab 1.2 mg/kg (N=35)
Anemia (Blood and lymphatic system disorders) | 2 | 17
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 13
Diarrhea (Gastrointestinal disorders) | 3 | 8
Oral mucositis (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 11
Vomiting (Gastrointestinal disorders) | 0 | 6
Chills (General disorders) | 0 | 3
Fatigue (General disorders) | 2 | 11
Fever (General disorders) | 1 | 3
Pain (General disorders) | 1 | 7
Mucosal infection (Infections and infestations) | 0 | 3
alanine aminotransferase increased (Investigations) | 2 | 6
Alkaline phosphatase increased (Investigations) | 3 | 7
Blood albumin increased (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 1 | 9
Neutrophil count decreased (Investigations) | 2 | 17
Platelet count decreased (Investigations) | 1 | 8
White blood cell decreased (Investigations) | 1 | 13
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia (Investigations) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Paresthesia (Nervous system disorders) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 16
Anxiety (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 6
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 3 | 4
Anal pain (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 2
Non-cardiac pain (General disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 5
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 1 | 0
Weight gain (Investigations) | 0 | 2
Weight loss (Investigations) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT01771107/Prot_SAP_000.pdf